CLINICAL TRIAL: NCT02989103
Title: Hyperthyroid Follow-Up Study
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917021; 17-C-N021
Record Dates: First submitted 2016-12-06; First posted 2016-12-12 (Estimated); Last update posted 2020-10-29 (Actual); Status verified 2020-10

CONDITIONS: All-Cause Mortality; Circulatory and Other Disease Mortality; Thyroid and Other Cancer Mortality
Keywords: Hyperthyroidism; Radiation; Mortality
MeSH Terms: conditions — Thyroid Diseases; Hyperthyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Hyperthyroidism Follow-up Cohort Study: Hyperthyroid patients enrolled and treated between 1946 and 1964 in 25 U.S. and 1 UK site

SUMMARY:
Background:

Hyperthyroidism is a common disease. It is very common for women. It is usually treated with Radioiodine (I-131). Some people think that this might cause cancer, even many years later. Past studies of people with hyperthyroidism have not been clear about cancer risks after I-131. Researchers want to look at a group of people with the disease who got I-131 many years ago. They want to look at how their health was months and years later.

Objective:

To learn more about disease risks in relation to radiation from I-131 treatment for hyperthyroidism.

Eligibility:

People who were part of the previous study. These are people who were diagnosed with hyperthyroidism at U.S. and U.K. hospitals from 1946 to 1964. About 95% of the participants have already died.

Design:

Researchers will examine data already collected by the past study. This includes data on participants later cancers and other health outcomes after they had I-131 treatment.

Researchers will compare that data to a National Death Index search.

This was already done for data up through 2003. This study will cover 2004 2014.

Researchers will not be in touch with study participants or their next of kin....

DETAILED DESCRIPTION:
Hyperthyroidism (thyrotoxicosis) is a relatively common disease, especially among women, and radioiodine (I-131) administration is the treatment of choice for most adult patients. There is concern about possible carcinogenic effects of I-131 therapy, but previous studies of hyperthyroid patients have not presented clear results regarding cancer risks following I-131 treatment. There also is public concern regarding late health consequences of I-131 exposure as this radioiodine is one of the primary release products from nuclear power generation and a principal component in fallout from nuclear power plant accidents. The Thyrotoxicosis Therapy Follow-up Study (TTFUS) cohort, assembled in 1961, comprises 35,000 subjects treated for hyperthyroidism at over 20 medical centers in the US and one in Great Britain between 1946 and 1964. This is among the largest group of hyperthyroid patients that has been followed up for subsequent cancer and other health outcomes. The proposed mortality follow-up study will enable us to assess nearly lifetime risk of cancer and other diseases in this unique cohort. Mortality follow-up data will extend the observation through 2015, adding 15 more years, via linkage with the National Death Index search. Recently estimated I-131 radiation doses to various body organs will allow refined dose response analysis, providing most definitive assessment of the nature and magnitude of the risk of cancer and other disease associated with I-131 exposure as well as end-results of I-131 and other treatment for hyperthyroidism.

ELIGIBILITY:
* INCLUSION:

Individuals treated for hyperthyroidism registered within the Thyrotoxicosis Therapy Follow-up Study (TTFUS) cohort that was assembled in 1961.

EXCLUSION:

Any individual that was NOT treated for hyperthyroidism registered within the Thyrotoxicosis Therapy Follow-up Study (TTFUS) cohort that was assembled in 1961.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort includes all hypothyroid patients treated with I-131, thyroid surgery, anti-thyroid drugs, or any combinations of these treatments between 1946 and 1964 at 25 U.S. and 1 UK institution. The cohort is largely female (79%), with a mean age at study entry (in 1961) of 46 years old. Hyperthyroidism patients in the cohort are classified as those with Graves disease (91%), toxic nodular goiter (8%), and unknown (1%).
Sampling Method: Non-Probability Sample
Enrollment: 35593 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
Cancer mortality rates | 1946 to 2014
  Mortality rates due to cancer in the cohort population.
Non-cancer mortality | 1946 to 2014
  Mortality rates due to non-cancer in the cohort population

CONTACTS AND LOCATIONS:
Overall Officials: Cari M Kitahara, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Social and Scientific Systems, Inc., Durham, North Carolina, United States

REFERENCES:
- [Background] Kitahara CM, Berrington de Gonzalez A, Bouville A, Brill AB, Doody MM, Melo DR, Simon SL, Sosa JA, Tulchinsky M, Villoing D, Preston DL. Association of Radioactive Iodine Treatment With Cancer Mortality in Patients With Hyperthyroidism. JAMA Intern Med. 2019 Aug 1;179(8):1034-1042. doi: 10.1001/jamainternmed.2019.0981. PMID 31260066
- [Background] Dobyns BM, Sheline GE, Workman JB, Tompkins EA, McConahey WM, Becker DV. Malignant and benign neoplasms of the thyroid in patients treated for hyperthyroidism: a report of the cooperative thyrotoxicosis therapy follow-up study. J Clin Endocrinol Metab. 1974 Jun;38(6):976-98. doi: 10.1210/jcem-38-6-976. No abstract available. PMID 4134013
- [Background] Ron E, Doody MM, Becker DV, Brill AB, Curtis RE, Goldman MB, Harris BS 3rd, Hoffman DA, McConahey WM, Maxon HR, Preston-Martin S, Warshauer ME, Wong FL, Boice JD Jr. Cancer mortality following treatment for adult hyperthyroidism. Cooperative Thyrotoxicosis Therapy Follow-up Study Group. JAMA. 1998 Jul 22-29;280(4):347-55. doi: 10.1001/jama.280.4.347. PMID 9686552